CLINICAL TRIAL: NCT06308302
Title: Comparative Effects of Inspiratory Muscle Training vs Expiratory Muscle Training Along With Aerobic Interval Training on Functional Performance and Fatigue Level in COPD Patients
Brief Title: Comparative Effects of IMT Vs EMT Along With AIT in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/RCR&AHS/23/0355
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: COPD
Keywords: Chronic Obstructive pulmonary disease; Dyspnea; Breathing Exercises; Pulmonary Disease; Fatigue; Functional Performance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Lung Diseases; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A (Inspiratory Muscles Training +Aerobic Interval Training)
  Interventions: Other: Group A (Inspiratory Muscles Training + Aerobic Interval Training)
- Group B (Experimental): Group B (Expiratory Muscles Training +Aerobic Interval Training)
  Interventions: Other: Group B (Expiratory Muscles Training +Aerobic Interval Training)

INTERVENTIONS:
Other: Group A (Inspiratory Muscles Training + Aerobic Interval Training) — Performed Inspiratory muscle training on a breather device (20), (10 inhales with maximum 3-sec hold), 3 sets with a 1-minute interval between each set, for 6 days a week along with aerobic interval training on alternate days (3 days a week for 20-25 minutes in 1st week, 30-35 minutes in 2nd week, 40 minutes in 3rd week, 45-60 minutes in 4th week each session). (120)
  Baseline treatment given is Aerobic interval training and COPD medications.
  Arms: Group A
Other: Group B (Expiratory Muscles Training +Aerobic Interval Training) — Performed Expiratory muscle training along with aerobic interval training on alternate days (3 days a week for 20-25 minutes in 1st week, 30-35 minutes in 2nd week, 40-45 minutes in 3rd week, 45-60 minutes in 4th week per session). (120)
  Baseline treatment given is Aerobic interval training and COPD medications.
  Arms: Group B

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is the 3rd leading cause of mortality and 7th leading cause of ill-health worldwide. It is characterized by persistent and progressive air flow resistance with expiratory flow more compromised as compared to inspiratory flow leading to CO2 retention and prominent hyperinflation of lungs. The overall effects of COPD on the patient's entire body include pulmonary, followed by extra-pulmonary manifestations in which musculoskeletal derangements are more pronounced and interfere with daily activities, further deteriorating the patient's health. Restricted air flow leads to an increase in shortness of breath on slight exertion and early fatigue or exhaustion of respiratory muscles due to over work. Literature from the past describes how COPD care has advanced and emphasizes the value of pulmonary rehabilitation in addition to medicinal management to treat decadence. Many studies show that Inspiratory muscle training has positive effect on ABG's, some PFT's and diaphragmatic function. Endurance and strength training improve patient activity of daily living and dyspnea.

This study intricate the collation of Respiratory Muscle Training and Aerobic Interval Training on functional performance, exertional dyspnea and fatigue level in patients diagnosed with COPD. A randomized controlled trial will be integrated with the sample size of 53 patients which is calculated through epi-tool. Age of selected Patients will fall between 30-55 years and will be randomly assigned into 2 groups. Group A (Experimental group A) will get Inspiratory breather training along-with Aerobic Interval Training, Group B (Experimental group B) will get Expiratory muscle training along-with Aerobic Interval Training (Same Protocol). Data will be gathered from Pulmonology wards and OPD of selected hospital. Clinical Assessment will be incorporated through Karnofsky performance scale, Fatigue Severity Scale, MmRC Dyspnea scale, Digital Spirometer, and 6MWT. Pre-intervention assessment measures and Post-intervention measures will be noted and results will be compared. Study Duration will be of 06 months after approval of synopsis. Data analysis will be done through SPSS.

Key words: Aerobic Interval training (AIT), The Breather Device (BD), 6-min walk test (6MWT), Fatigue severity scale (FSS), Modified Medical Research Council dyspnea scale (mMRC), Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosed case of COPD.
* Participants must be between the ages of 30 and 55 years old.
* Participants must have GOLD II and III stage COPD.
* Both men and women are eligible for the study.

Exclusion Criteria:

* Participants with a history of cardiovascular disease.
* Participants with a history of neurological disease.
* Participants with a history of orthopaedic disease.
* Participants with a history of neuromuscular disease.
* Participants who had experienced a recent COPD exacerbation within the past 3 months.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Modified Medical Research Council (mMRC) Dyspnea Scale | 4 Weeks
  A widely recognized tool for evaluating the level of breathlessness experienced by patients with COPD. It provides a simple and efficient method of assessing the baseline functional disability due to dyspnea. experiencing breathlessness with strenuous exercise.
  The scale ranges from 0 to 4, with each grade representing a different level of breathlessness, from only experiencing breathlessness with strenuous exercise (Grade 0) to being too breathless to leave the house or experiencing breathlessness when dressing or undressing (Grade 4).
6 Minute Walk Test | 4 Weeks
  The 6-Minute Walk Test (6MWT) is a sub-maximal exercise test used to assess aerobic capacity and endurance, particularly in patients with COPD. The score of the 6MWT is the distance a patient walks in 6 minutes. The patient may take as many standing rests as they like, but the timer should keep going. The 6MWT measures exercise tolerance in people with various health conditions.
Karnofsky Performance Scale (KPS) | 4 Weeks
  The Karnofsky Performance Scale (KPS) is an assessment tool used to predict the length of survival in terminally ill patients.It's an 11-point rating scale ranging from normal functioning (100) to dead (0) in ten-point increments. The higher the score, the more independent the person is.
Fatigue Severity Scale (FSS) | 4 week
  A tool used to measure the severity of fatigue in patients with Chronic Obstructive Pulmonary Disease (COPD). It's a 9-item questionnaire where each item is scored on a 7-point scale, with 1 indicating strong disagreement and 7 indicating strong agreement. The total score ranges from 9 to 63, with higher scores indicating greater fatigue severity.
FEV1 | 4 Weeks
  A Digital Spirometer is a device used to measure the volume and speed of air a person can inhale and exhale. It is often used to diagnose and monitor conditions like COPD. The spirometer measures the Forced Expiratory Volume in 1 second (FEV1), which is how much air you can exhale in the first second after a full inhalation. The FEV1 and FVC values are used to diagnose conditions like COPD.
FVC | 4 weeks
  Digital Spirometer will be used to measure the volume and speed of air a person can inhale and exhale. The spirometer measures the Forced Vital Capacity (FVC), which is the largest amount of air that you can forcefully exhale after breathing in as deeply as you can. Pre-post reading will be taken. it is measures in liters.
FEV1/FVC | 4 weeks
  Digital Spirometer is a device used to measure the volume and speed of air a person can inhale and exhale. The FEV1 and FVC values are used to diagnose conditions like COPD. The ratio of FEV1 to FVC (FEV1/FVC) is calculated and expressed as a percentage. Pre-Post readings will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSCPPT, Principal Investigator — Ripha International University-LHR
Locations (1):
- Al-Zahra Rehabilitation Center, Gulab Devi Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adeloye D, Song P, Zhu Y, Campbell H, Sheikh A, Rudan I; NIHR RESPIRE Global Respiratory Health Unit. Global, regional, and national prevalence of, and risk factors for, chronic obstructive pulmonary disease (COPD) in 2019: a systematic review and modelling analysis. Lancet Respir Med. 2022 May;10(5):447-458. doi: 10.1016/S2213-2600(21)00511-7. Epub 2022 Mar 10. PMID 35279265
- [Background] Landt E, Colak Y, Lange P, Laursen LC, Nordestgaard BG, Dahl M. Chronic Cough in Individuals With COPD: A Population-Based Cohort Study. Chest. 2020 Jun;157(6):1446-1454. doi: 10.1016/j.chest.2019.12.038. Epub 2020 Jan 25. PMID 31987882
- [Background] Gutierrez Villegas C, Paz-Zulueta M, Herrero-Montes M, Paras-Bravo P, Madrazo Perez M. Cost analysis of chronic obstructive pulmonary disease (COPD): a systematic review. Health Econ Rev. 2021 Aug 17;11(1):31. doi: 10.1186/s13561-021-00329-9. PMID 34403023
- [Background] Chen S, Kuhn M, Prettner K, Yu F, Yang T, Barnighausen T, Bloom DE, Wang C. The global economic burden of chronic obstructive pulmonary disease for 204 countries and territories in 2020-50: a health-augmented macroeconomic modelling study. Lancet Glob Health. 2023 Aug;11(8):e1183-e1193. doi: 10.1016/S2214-109X(23)00217-6. PMID 37474226
- [Background] Agarwal D. COPD generates substantial cost for health systems. Lancet Glob Health. 2023 Aug;11(8):e1138-e1139. doi: 10.1016/S2214-109X(23)00304-2. No abstract available. PMID 37474208
- [Background] Carter P, Lagan J, Fortune C, Bhatt DL, Vestbo J, Niven R, Chaudhuri N, Schelbert EB, Potluri R, Miller CA. Association of Cardiovascular Disease With Respiratory Disease. J Am Coll Cardiol. 2019 May 7;73(17):2166-2177. doi: 10.1016/j.jacc.2018.11.063. Epub 2019 Mar 4. PMID 30846341
- [Background] Hughes MJ, McGettrick HM, Sapey E. Shared mechanisms of multimorbidity in COPD, atherosclerosis and type-2 diabetes: the neutrophil as a potential inflammatory target. Eur Respir Rev. 2020 Mar 20;29(155):190102. doi: 10.1183/16000617.0102-2019. Print 2020 Mar 31. PMID 32198215
- [Background] Li Y, Gao H, Zhao L, Wang J. Osteoporosis in COPD patients: Risk factors and pulmonary rehabilitation. Clin Respir J. 2022 Jul;16(7):487-496. doi: 10.1111/crj.13514. Epub 2022 Jun 10. PMID 35688435
- [Background] Li Z, Liu S, Wang L, Smith L. Mind-Body Exercise for Anxiety and Depression in COPD Patients: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2019 Dec 18;17(1):22. doi: 10.3390/ijerph17010022. PMID 31861418
- [Background] Zou M, Zhang W, Xu Y, Zhu Y. Relationship Between COPD and GERD: A Bibliometrics Analysis. Int J Chron Obstruct Pulmon Dis. 2022 Dec 6;17:3045-3059. doi: 10.2147/COPD.S391878. eCollection 2022. PMID 36510485